CLINICAL TRIAL: NCT01235026
Title: Impact of the Administration of a Synbiotic on Low Grade Inflammation in Obese Subjects
Brief Title: Synbiotics and Low Grade Inflammation in Obese Subjects
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Chile (Other)
Responsible Party: Martin Gotteland, University of Chile
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: Fondecyt-1080519
Record Dates: First submitted 2010-11-01; First posted 2010-11-05 (Estimated); Last update posted 2010-12-17 (Estimated); Status verified 2010-10

CONDITIONS: Obesity; Diabetes Mellitus Type-2; Insulin Resistance; Metabolic Syndrome
Keywords: Obesity; Type-2 Diabetes; Metabolic syndrome; Low grade inflammation; Metabolic endotoxinemia; Insulin resistance; Lipopolysaccharide; LPS-binding protein; sCD14; Synbiotic; Oligofructose; Bifidobacterium animalis subsp. lactis Bb12; probiotic; Prebiotic
MeSH Terms: conditions — Obesity; Insulin Resistance; Metabolic Syndrome | interventions — Synbiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Synbiotic (Experimental): Dietary Supplement: Synbiotic: combination of the prebiotic "Oligofructose" with the probiotic "Bifidobacterium animalis subsp. lactis Bb12"
  Interventions: Dietary Supplement: Synbiotic
- Placebo (Placebo Comparator): Dietary supplement: placebo: maltodextrin
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Synbiotic — 5g of the prebiotic "Oligofructose" + 1 g of the probiotic "Bifidobacterium animalis subsp. lactis Bb12" (4x10^10 CFU/g), twice a day, for 6 weeks.
  Arms: Synbiotic
Dietary Supplement: Placebo — 6g of maltodextrin, twice a day for 6 weeks.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether the daily administration of a synbiotic (oligofructose and Bifidobacterium animalis subsp. lactis Bb12) for six weeks contributes to improve the glucose tolerance and the low grade inflammation (as reflected as the plasmatic concentrations of ultrasensitive CRP, IL-6, sCD14 and LPS-binding protein) in obese subjects.

DETAILED DESCRIPTION:
Obesity is associated with a spectrum of metabolic disorders including high blood pressure, dyslipidemia, insulin resistance and a state of low grade inflammation that predispose individuals to the development of type-2 diabetes mellitus and cardiovascular diseases. The intestinal microbiota has been recently proposed as a new actor in the development of obesity and its complications. In animal models, high-fat diets have been shown to affect the intestinal microbiota, increasing colonic gram-negative bacteria and lipopolysaccharide (LPS) concentrations, resulting in an impaired gastrointestinal barrier function and in subsequent endotoxinemia in the animals. This phenomenon would trigger chronic inflammatory and metabolic disorders leading to insulin resistance and other complication such as hepatic steatosis. Probiotics and prebiotics are GRAS (Generally recognized as safe) food ingredients which have been proposed to maintain the balance of the intestinal microbiota. Studies in mice fed a high fat diet have shown that the administration of oligofructose increases the counts of Bifidobacterium spp. in the colon and correlatively induced decreases of the endotoxinemia and low-grade inflammation while at the same time improving insulin sensitivity.

On the basis of these antecedents, the aim of this study is to determine whether the intake of a synbiotic product (B. animalis subsp. lactis BB12+ Oligofructose) for six weeks contributes to improve the low grade inflammation and glucose tolerance of obese subjects.

Obese subjects will be randomized into two groups (Synbiotic or Placebo) stratifying by sex and age. Anthropometric data (body composition by Bod-pod, weight, height, waist circumference) and systolic and diastolic blood pressure will be registered. A food survey will be carried out by a trained dietitian to quantify fat consumption. Each subject of the Synbiotic group must ingest one gram of BB12 (containing 1010 CFU) and 5 g of oligofructose twice a day for 6 weeks while those from the Control group will receive the corresponding placebo (maltodextrin). Digestive symptoms as well as stool frequency and consistency will be registered daily during the study using ad hoc forms and the Bristol Chart.

Blood samples will be obtained at baseline, at the end of the six weeks period and one month after the end of the treatment, to determine lipid profiles and ultrasensitive C-reactive protein (CRP); plasmatic biomarkers of inflammation including IL-6, LPS binding protein and sCD14 will be also determined by Elisa using commercial kits. At the same times, a glycemia /insulinemia curve will be performed in the fasted subjects, as well as an intestinal permeability test (lactulose/mannitol/sucralose) to assess their gut barrier function. A fresh stool sample will be also obtained to characterize some bacterial population of their IM (Bifidobacterium, Lactobacillus, F. prausnitzii, Bacteroides and Clostridium cluster) by real-time PCR.

ELIGIBILITY:
Inclusion Criteria:

* BMI > 30
* Non-smokers

Exclusion Criteria:

* Current digestive diseases or antecedents of chronic digestive diseases and/or malabsorption (celiac disease, Inflammatory bowel diseases, gastroduodenal ulcers, digestive malignancies, etc)
* Use of drugs that could interfere with the intestinal microbiota or with the integrity of the gut barrier function (antibiotics, anti-inflammatory drugs, laxatives, prokinetics, etc.) during the three weeks preceding the start the study
* Treatments (medication or nutritional program) affecting body weight or glucose control
* Basal glycemia>130mg/dl (evaluated with glucose-meter)
* Immunodeficiencies (HIV, chemotherapy, radiotherapy, organ transplant).
* Current participation or recent previous having participation in another clinical trial.
* Pregnant or breastfeeding women.
* Consumption of probiotic products
* Drug or alcohol abuse

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Estimated)
Dates: Start 2010-11; Primary Completion 2010-12 (Estimated); Study Completion 2011-01 (Estimated)

PRIMARY OUTCOMES:
Plasmatic Interleukin-6 (IL-6) | 6 weeks
  Plasmatic IL-6 will be determined after 6 weeks of administration of the synbiotic and compared with the IL-6 values at baseline.

SECONDARY OUTCOMES:
Plasmatic LPS-binding protein | 6 weeks
  Plasmatic LPS-binding protein (LBP) will be determined after 6 weeks of administration of the synbiotic and compared with the LBP values at baseline.
Plasmatic sCD14 | 6 weeks
  Plasmatic sCD14 will be determined after 6 weeks of administration of the synbiotic and compared with the sCD14 values at baseline.
glucose tolerance curve | 6 weeks
  Glucose tolerance will be determined after 6 weeks of administration of the synbiotic and compared with glucose tolerance at baseline.
Lipid profile | 6 weeks
  Lipid profile will be determined after 6 weeks of administration of the synbiotic and compared with the lipid profile at baseline.
plasmatic ultrasensitive C-Reactive Protein | 6 weeks
  Plasmatic ultrasensitive CRP will be determined after 6 weeks of administration of the synbiotic and compared with the usCRP values at baseline.
Plasmatic IL-6 | 10 weeks
  Plasmatic IL-6 will be determined after a 1-month washout period without synbiotic administration (week 10)and compared with the baseline and post-treatment (6 weeks) values.
Plasmatic LBP | 10 weeks
  Plasmatic LBP will be determined after a 1-month washout period without synbiotic administration (week 10)and compared with the baseline and post-treatment (6 weeks) values.
Plasmatic sCD14 | 10 weeks
  Plasmatic sCD14 will be determined after a 1-month washout period without synbiotic administration (week 10)and compared with the baseline and post-treatment (6 weeks) values.
Glucose tolerance curve | 10 weeks
  Glucose tolerance curves will be determined after a 1-month washout period without synbiotic administration (week 10)and compared with the baseline and post-treatment (6 weeks) values.
Lipid profile | 10 weeks
  Lipid profile will be determined after a 1-month washout period without synbiotic administration (week 10)and compared with the baseline and post-treatment (6 weeks) values.
Plasmatic usCRP | 10 weeks
  Plasmatic usCRP will be determined after a 1-month washout period without synbiotic administration (week 10)and compared with the baseline and post-treatment (6 weeks) values.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Nutrition and Food Technology (INTA), University of Chile, Santiago, Chile

REFERENCES:
- [Background] Cani PD, Bibiloni R, Knauf C, Waget A, Neyrinck AM, Delzenne NM, Burcelin R. Changes in gut microbiota control metabolic endotoxemia-induced inflammation in high-fat diet-induced obesity and diabetes in mice. Diabetes. 2008 Jun;57(6):1470-81. doi: 10.2337/db07-1403. Epub 2008 Feb 27. PMID 18305141
- [Background] Cani PD, Neyrinck AM, Fava F, Knauf C, Burcelin RG, Tuohy KM, Gibson GR, Delzenne NM. Selective increases of bifidobacteria in gut microflora improve high-fat-diet-induced diabetes in mice through a mechanism associated with endotoxaemia. Diabetologia. 2007 Nov;50(11):2374-83. doi: 10.1007/s00125-007-0791-0. Epub 2007 Sep 6. PMID 17823788
- [Background] Ley RE, Turnbaugh PJ, Klein S, Gordon JI. Microbial ecology: human gut microbes associated with obesity. Nature. 2006 Dec 21;444(7122):1022-3. doi: 10.1038/4441022a. PMID 17183309
- [Background] Wright SD, Ramos RA, Tobias PS, Ulevitch RJ, Mathison JC. CD14, a receptor for complexes of lipopolysaccharide (LPS) and LPS binding protein. Science. 1990 Sep 21;249(4975):1431-3. doi: 10.1126/science.1698311.
- [Background] Brunser O, Figueroa G, Gotteland M, Haschke-Becher E, Magliola C, Rochat F, Cruchet S, Palframan R, Gibson G, Chauffard F, Haschke F. Effects of probiotic or prebiotic supplemented milk formulas on fecal microbiota composition of infants. Asia Pac J Clin Nutr. 2006;15(3):368-76. PMID 16837430